CLINICAL TRIAL: NCT04848519
Title: Immune Checkpoint Inhibitors With or Without Propranolol Hydrochloride In Patients With Urothelial Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jacqueline Brown, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002186; NCI-2021-00437 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); WINSHIP5200-20 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Locally Advanced Bladder Urothelial Carcinoma; Locally Advanced Renal Pelvis Urothelial Carcinoma; Locally Advanced Ureter Urothelial Carcinoma; Locally Advanced Urethral Urothelial Carcinoma; Locally Advanced Urothelial Carcinoma; Metastatic Bladder Urothelial Carcinoma; Metastatic Renal Pelvis Urothelial Carcinoma; Metastatic Ureter Urothelial Carcinoma; Metastatic Urethral Urothelial Carcinoma; Metastatic Urothelial Carcinoma; Stage IV Bladder Cancer AJCC v8; Stage IV Renal Pelvis Cancer AJCC v8; Stage IV Ureter Cancer AJCC v8; Stage IV Urethral Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms | interventions — pembrolizumab; Propranolol; Nivolumab; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (propranolol hydrochloride, immune checkpoint inhibitor) (Experimental): The specific ICI that the subject would receive will be dependent on the clinical need and associated FDA approval.
  Interventions: Drug: Pembrolizumab; Drug: Propranolol Hydrochloride; Drug: Nivolumab; Drug: Avelumab
- Treatment (immune checkpoint inhibitor) (Other): The specific ICI that the subject would receive will be dependent on the clinical need and associated FDA approval.
  Interventions: Drug: Pembrolizumab; Drug: Nivolumab; Drug: Avelumab

INTERVENTIONS:
Drug: Pembrolizumab — Given IV as first line for locally advanced or metastatic urothelial carcinoma who are not eligible for platinum-based chemotherapy; or second line for locally advanced or metastatic urothelial carcinoma after progression on platinum-based chemotherapy
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Propranolol Hydrochloride — Given PO for patients on the ICI plus propranolol arm
  Other Names: Inderal
  Arms: Treatment (propranolol hydrochloride, immune checkpoint inhibitor)
Drug: Nivolumab — Given IV as adjuvant treatment of urothelial carcinoma in high risk of disease recurrence after undergoing radical resection
Drug: Avelumab — Given IV as maintenance treatment in locally advanced or metastatic urothelial carcinoma following no progression on first-line platinum-containing chemotherapy

SUMMARY:
This research study is an open label study designed to evaluate the safety and translational correlative changes of the combination of propranolol hydrochloride and immune checkpoint inhibitors (ICI) in subjects with urothelial carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety of the combination of propranolol hydrochloride and immune checkpoint inhibitors in urothelial cancer as measured by the incidence of adverse events according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0

SECONDARY OBJECTIVE:

I. To describe response and survival outcomes for ICI plus or minus propranolol in patients with urothelial cancer as measured by ORR per RECIST 1.1 (only for subjects receiving avelumab and pembrolizumab as ICI), profession free survival (PFS) and overall survival (OS).

TERTIARY/EXPLORATORY OBJECTIVE:

I. To measure overall response rate (ORR) along with correlative changes in peripheral T-cell subsets, myeloid derived suppressor cells (MDSC), blood inflammatory markers and blood cytokines before and after treatment for patients receiving ICI plus propranolol vs. ICI alone. Available archival tissue will also be collected for tissue-based assays.

OUTLINE:

Patients who meet eligibility criteria and consent for enrollment in the trial will be on one of the two study cohorts. Assignment to cohorts will be sequentially, in a 1:1 fashion, starting with the ICI plus propranolol cohort. The specific ICI that the subject would receive will be dependent on the clinical need and associated FDA approval.

ICI PLUS PROPRANOLOL COHORT:

1. Propranolol: Participants will remain on propranolol 30mg twice daily for the duration of the trial unless unacceptable toxicity or withdrawal of consent. Patients who develop toxicity and stop propranolol will remain on trial for endpoint measurement.

PLUS

Pembrolizumab: Participants will receive 200mg IV on Day 1, every 3 weeks. Pembrolizumab would be continued for up to 2 years in the absence of disease progression or unacceptable toxicity.

OR

Avelumab: Participants will receive Avelumab at a dose of 10 mg per kilogram of body weight, IV on Day 1 every 2 weeks until disease progression or unacceptable toxicity.

OR

Nivolumab: Participants will receive Nivolumab (480mg) IV on every 4 weeks for up to 1 year or until disease recurrence or discontinuation from the trial.

ICI ALONE COHORT:

Pembrolizumab: Participants will receive 200mg IV on Day 1, every 3 weeks. Pembrolizumab would be continued for up to 2 years in the absence of disease progression or unacceptable toxicity.

OR

Avelumab: Participants will receive Avelumab at a dose of 10 mg per kilogram of body weight, IV on Day 1 every 2 weeks until disease progression or unacceptable toxicity

OR

Nivolumab: Participants will receive Nivolumab (480mg) IV on every 4 weeks for up to 1 year or until disease recurrence or discontinuation from the trial.

After completion of study treatment, patients are followed up at 30 days, then every 12 weeks for up to 2 years.

ELIGIBILITY:
INCLUSION CRITERIA

1. Male or Female
2. Age ≥18 years
3. ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
4. Patients must have histologically confirmed urothelial carcinoma planned for treatment with any of the following at the genitourinary oncology clinics of Emory University's Winship Cancer Institute under the list FDA approved indications:

   * Pembrolizumab: first line for locally advanced or metastatic urothelial carcinoma who are not eligible for platinum-based chemotherapy; or second line for locally advanced or metastatic urothelial carcinoma after progression on platinum-based chemotherapy)
   * Avelumab: maintenance treatment in locally advanced or metastatic urothelial carcinoma following no progression on first-line platinum-containing chemotherapy
   * Nivolumab: adjuvant treatment of urothelial carcinoma in high risk of disease recurrence after undergoing radical resection. High risk disease as defined in Checkmate 274: pathological stage of pT3, pT4a, or pN+ and patient not eligible for or declined adjuvant cisplatin-based combination chemotherapy for patients who had not received neoadjuvant cisplatin-based chemotherapy and pathological stage of ypT2 to ypT4a or ypN+ for patients who received neoadjuvant cisplatin
5. Patients must have adequate organ and marrow function, within 28 days of Cycle 1 Day 1, at the discretion of the investigator.
6. The effects of study drugs on the developing human fetus are unknown. For this reason, female of child-bearing potential (FCBP) must have a negative serum or urine pregnancy test prior to starting therapy.
7. FCBP and men treated or enrolled on this protocol must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 3 months after completion of study drug administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

   - A female of childbearing potential (FCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
8. Completion of all previous therapy (including surgery, radiotherapy, chemotherapy, immunotherapy, or investigational therapy) for the treatment of cancer ≥ 4 weeks before the start of study therapy.
9. Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification (Appendix B). To be eligible for this trial, patients should be class IIB or better.

   * Patients without existing cardiac disease that raise the risk of complications who consent for the trial will proceed with trial participation.
   * Patients with existing cardiac disease that could raise the risk of complications will be referred at the discretion of the investigator to a cardio-oncologist who is a co-investigator on the trial (or general cardiologist) for cardiac optimization prior to starting propranolol.
10. Life expectancy > 12 weeks as determined by the Investigator.
11. Willingness and ability of the subject to comply with scheduled visits, drug administration plan, protocol-specified laboratory tests, other study procedures, and study restrictions.
12. Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation.

EXCLUSION CRITERIA

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier (i.e., have residual toxicities > Grade 2).
2. Patients who are receiving any other investigational agents or an investigational device within 21 days before administration of first dose of study drugs.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the agents used in study.
4. Contraindication to ICI per investigator discretion.
5. Uncontrolled current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Significant cardiovascular disease (e.g., myocardial infarction, arterial thromboembolism, cerebrovascular thromboembolism) within 3 months prior to start of study therapy; angina requiring therapy; symptomatic peripheral vascular disease; New York Heart Association Class 3 or 4 congestive heart failure; or uncontrolled Grade ≥3 hypertension (diastolic blood pressure ≥100 mmHg or systolic blood pressure ≥160 mmHg) despite antihypertensive therapy.
7. Contraindication to a beta blocker: cardiac conditions that significantly raise the risk of cardiopulmonary complications, including unstable angina, uncontrolled heart failure, symptomatic bradycardia, and severe asthma.
8. Current use of an oral or intravenous beta blocker (e.g. atenolol, bisoprolol, carvedilol, labetalol, metoprolol, nadolol, sotalol, among other beta blockers) with inability to safely switch to a non-beta blocker agent. The washout for current users should be at least 14 days with enough transition period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 2 years
  Assessed according to the Common Terminology Criteria for Adverse Events version 5.0. Descriptive statistics will be used to summarize the toxicity profile of the intervention. Toxicities will be tabulated by grade, association, and cycle number.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 2 years
  Kaplan-Meier methods will be used to estimate median survival time or time-specific survival rate with 95% confidence interval for PFS.
Overall survival (OS) | 2 years
  Kaplan-Meier methods will be used to estimate median survival time or time-specific survival rate with 95% confidence interval for OS.
Objective Response Rate (ORR) | 2 years
  Defined as the proportion of subjects only receiving avelumab and pembrolizumab as ICI.

OTHER OUTCOMES:
Immune profile and changes in selected biomarkers and cell subsets | 2 years
  Correlative changes in peripheral T-cell subsets, myeloid derived suppressor cells, blood inflammatory markers and blood cytokines before and after treatment, will first be described by summary statistics. Descriptive statistics on continuous data will include mean, median, standard deviation, and range (as well as geometric means and geometric coefficient of variation for pharmacokinetic parameters), while categorical data will be summarized using frequency counts and percentages. Graphical summaries of the data may be presented. Their correlation with clinical efficacy endpoints will be carried out by logistic regression model for ORR or Cox proportional hazard mode for time to even outcomes (OS or PFS).

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Brown, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT04848519/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT04848519/ICF_001.pdf